CLINICAL TRIAL: NCT05118880
Title: Evaluation Of The Effectiveness Of The Peer Bullying Consultancy Program Based On The Interpersonal Relations Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kadriye Demir (Other Government)
Responsible Party: Sponsor-Investigator, Kadriye Demir, Assistant Prof., Lokman Hekim University
Organization: Lokman Hekim University (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LokmanHekimU-SBF-HB-KD-01
Record Dates: First submitted 2021-10-01; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Perr Bulling, Middle School Child, School Nursing, Peplau-Interpersonel Relationship Theory
Keywords: Peer Bullying; Consultancy Program; Nurse, Interpersonal Relations; Model; Peblau

STUDY DESIGN:
Intervention Model Description: The research was conducted in the pretest-posttest experimental research design with intervention-control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): the children enrolled in the Peer Bullying Counseling Program based on the Interpersonal Relationship Model
  Interventions: Other: Peer Bullying Counseling Program based on the Interpersonal Relationship Model
- control group (No Intervention)

INTERVENTIONS:
Other: Peer Bullying Counseling Program based on the Interpersonal Relationship Model — The content of the program was created by the researcher in line with the issues that peer bullying children need support based on their bullying-related characteristics in the light of the relevant literature. Education topics prepared in this framework; 'Empathy', 'Peer Bullying', 'Anger Management' and 'Happy Friendship Relationships' were determined. The main nursing problem of the research is "peer bullying". The main purpose of the Peer Bullying Counseling Program is to improve the empathy skills of the bullying child, to enable them to gain the right perspective towards bullying, to develop anger control, and to help them establish happy friendships. The content of the Peer Bullying Counseling Program; drawing, brainstorming, empathy demonstration, white paper activity, educational matching game, peer bullying demonstration, case studies, educational emotion puzzle game, anger control information video were applied using educational techniques.
  Arms: İntervention group

SUMMARY:
The research was conducted in experimental design with intervention-control group and pretest-posttest in order to examine the effectiveness of the Peer Bullying Consultancy Program (PBCP), is based on the Interpersonal Relations Model (IPM), on 11-12 years old children who are bullying. The sample group of the study consisted of children (intervention group/n=29; control group/n=32) were attending 5th and 6th grades in two different randomized designated secondary schools after stratified sampling, had high Peer Bullying Determination Scale Bully Behavior. The PBCP was implemented to the children in the intervention group in 2 face-to-face and 5 online individual interviews in 26 days. To increase the peer bullying cognition level, to develop empathy skills, to improve friendship relations, to increase anger control of children who are bullying in intervention group, content suitable for age characteristics was developed within the scope of PBCP various training techniques (brainstorming, educational game, demonstration, case study, video watching) used. The data were collected using Sociodemographic Information Form, the Bullying Related Cognitions Scale for Children (BRCSC), the Empathy Scale for Children and Adolescents (ESCA), Friendship Relations and Anger Control Assessment Form. Data collection tools were applied to the children in the intervention group at the beginning and at the end of the PBCP, and to the children in the control group with an interval of 26 days. In the study, children in the intervention group had lower scores on the BRCSC; had higher scores on the ESCA, Self-Reporting Happiness Level in Friendship Relations, Sample Behavior Knowledge Level for Happy Friendship, Understanding Level of Anger Symtoms, Knowledge Level of Anger Control and Self-Reporting Anger Control Level than the children in the control group (p<0.05). It has been determined the PBCP based on the IRM is effective for children aged 11-12 who are bullying. It is recommended nurses develop model-based, individual counseling and training program in which different educational techniques are used in accordance with the age characteristics in order to support the growth, development of children who are bullying within the framework of their roles such as advocate, consultant, leader.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion in the study are as follows.

  * Being 11 or 12 years old,
  * Having an internet connection at home,
  * Having a computer and/or phone for internet access,
  * Having at least one standard deviation above the school average in the PBIS-SSB sub-dimension score,
  * The voluntary acceptance of the child and his/her parents to participate in the research

Exclusion Criteria:

• Having any physical or mental health problems,

. Having a diagnosis of chronic disease

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2021-01-24 (Actual)

PRIMARY OUTCOMES:
Bullying Cognitions Scale for Children mean scores (BCSC) | Pre-test and post-test
  The BCSC was developed to assess the cognitive characteristics associated with peer bullying in children. The twenty-two-item scale was graded in a 4-point likert type ('completely true', 'quite true', 'somewhat true', 'not true at all'). The 'completely correct' response was rated as 4 points, the 'quite correct' response as 3 points, the 'somewhat correct' response as 2 points, and the 'not at all correct' response as 1 point. There is no reverse item in the scale. The scale is evaluated with a total score. The highest total score that can be obtained from the scale is "88" and the lowest score is "22". The higher the scores, the higher the cognitions about bullying. In other words, bullying is considered normal and normal.
Empathy Scale for Children and Adolescents (ESCA) | Pre-test and post-test
  The scale consists of 21 items. The scale is filled by giving one of the two answers as 'Yes' or 'No' to its items. The 'Yes' response was scored as 1 point, and the 'No' response as 0 points. However, some items (2,8,9,14,15,16,17,19,20 and 21) in the scale are reverse scored. In this case, 1 point was given to the "no" answer given to the item in question, and 0 point was given to the "yes" answer. The lowest score that can be obtained from the scale is 0, and the highest score is 21. As the score obtained from the scale increases, the empathic tendency increases, and as the score decreases, the empathic tendency decreases. The internal consistency coefficient of the scale was found to be 0.84 by Gürtunca and Karakale.

SECONDARY OUTCOMES:
Friendship Relations and Anger Control Evaluation Form (FRACEF) | Pre-test and post-test
  The Friendship Relations and Anger Control Evaluation Form was created considering the PBCP (Peer Bullying Counseling Program) content. The form was prepared to measure the happiness levels of children in friendship relationships, sample behavior information about happy friendship relationships, and their knowledge and competence levels about anger control. The Friendship Relations and Anger Control Evaluation Form consists of 5 questions, two for happy friendship relationships and three for anger control. A total of 50 points can be obtained from the form, with 10 points for each question.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadriye Demir, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
SPSS data will be shared during the publication of the article in accordance with the principle of protection of personal data.
  Evaluation of Data:
  Evaluation of the data was made in SPSS for Windows 11.5 (Chicago INC.) package program. Number, percentage, arithmetic mean, standard deviation, median, and minimum-maximum values were used in the intra-group distribution of descriptive data and scale scores. Non-parametric tests (Wilcoxon Test for intragroup difference, Man-Whitney U Test for intergroup difference) were used for statistical analysis of data that did not show normal distribution. The Kolmogorov-Smirnov test was used in the control group with an n≥30 score for the normal distribution of the scale mean scores. Statistical significance value was accepted as p<0.05.
  It is aimed that this research will be published in the Journal of School Nursing.